CLINICAL TRIAL: NCT05137119
Title: Staphylococcus Aureus Network Adaptive Platform Trial
Acronym: SNAP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Berry Consultants (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Menzies School of Health Research (Other); Aotearoa Clinical Trials (Unknown); Queensland University of Technology (Other); Sunnybrook Health Sciences Centre (Other); Tan Tock Seng Hospital (Other); Telethon Kids Institute (Other); The Peter Doherty Institute for Infection and Immunity (Other); The University of Queensland (Other); UMC Utrecht (Other); Radboud University Medical Center (Other); King's College London (Other); Rambam Health Care Campus (Other); University College, London (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CT19029
Record Dates: First submitted 2021-04-25; First posted 2021-11-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-07

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: Methicillin-resistant Staphylococcus aureus (MRSA); Methicillin-susceptible Staphylococcus aureus (MSSA); Penicillin-susceptible Staphylococcus aureus (PSSA); Staphylococcus aureus; S. aureus; Staph Aureus Bacteremia (SAB)
MeSH Terms: conditions — Staphylococcal Infections | interventions — Cefazolin; Penicillins; Penicillin G; Clindamycin; Lincomycin; Vancomycin; Daptomycin

STUDY DESIGN:
Intervention Model Description: Participants enrolled into the study have the option of deciding whether to be randomised in one or more (if available) treatment domains concurrently, if they meet the eligibility criteria.
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Methicillin-resistant staphylococcus aureus (MRSA) - Standard Therapy Arm (backbone therapy) (No Intervention): Vancomycin or Daptomycin - Standard Therapy Arm
  Either intravenous vancomycin dosed as per Australian Therapeutic Guidelines: This includes a loading dose of 25 mg/kg (up to 3000mg) if considered appropriate by the treating clinician, initial maintenance dosing at 15-20 mg/kg q12h, with subsequent adjustment to maintain area under the concentration-time curve (AUC) of 400 to 600 mg.hr/L OR trough levels at 10-20 mg/L, and the initial level taken 48-72 hours after the initiation of the first dose. Daptomycin 8-10mg/kg per day intravenously. The choice of vancomycin or daptomycin will be at the clinician's discretion. Dosing will be based on renal function.
- Methicillin-resistant staphylococcus aureus (MRSA) - Standard + B-Lactam Arm (backbone therapy) (Experimental): Vancomycin or Daptomycin (Standard Therapy) + Beta-Lactam (β-lactam) Arm
  In addition to standard treatment an intravenous β-lactam will be added for the first 7 calendar days following randomisation (day 1 being the day of randomisation - hence patients will receive 6-7 days of β-lactam). This β-lactam will be intravenous cefazolin 2g every 8 hours. For patients with renal impairment the intravenous cefazolin administration doses will be adjusted.
  Interventions: Drug: Cefazolin; Drug: Vancomycin
- Methicillin-susceptible staphylococcus aureus (MSSA) - Standard Therapy Arm (backbone therapy) (No Intervention): Flucloxacillin or cloxacillin - Standard Therapy Arm
  Either intravenous flucloxacillin/cloxacillin 2g every 4 or 6 hours. The minimum protocol duration of allocated study treatment is 14 days for those not allocated to early oral switch, and 5 days for those allocated to early oral switch. For patients with renal impairment or critical illness the intravenous flucloxacillin administration dose will be adjusted.
- Methicillin-susceptible staphylococcus aureus (MSSA) - Interventional Arm (backbone therapy) (Experimental): Cefazolin - Interventional Arm
  Intravenous cefazolin 2g every 6 or 8 hours. The minimum protocol duration of allocated study treatment is 14 days for those not allocated to early oral switch, and 5 days for those allocated to early oral switch. For patients with renal impairment or critical illness the intravenous cefazolin administration dose will be adjusted.
  Interventions: Drug: Cefazolin
- Penicillin-susceptible staphylococcus aureus (PSSA) - Standard Therapy Arm (backbone therapy) (No Intervention): Flucloxacillin or cloxacillin - Standard Therapy Arm
  Either intravenous flucloxacillin/cloxacillin 2g every 4 or 6 hours. The minimum protocol duration of allocated study treatment is 14 days for those not allocated to early oral switch, and 5 days for those allocated to early oral switch. For patients with renal impairment or critical illness the intravenous flucloxacillin administration dose will be adjusted.
- Penicillin-susceptible staphylococcus aureus (PSSA) - Interventional Arm (backbone therapy) (Experimental): Benzylpenicillin - Interventional Arm
  Intravenous benzylpenicillin 1.8g (3 million units) every 4 or 6 hours. The minimum protocol duration of allocated study treatment is 14 days for those not allocated to early oral switch, and 5 days for those allocated to early oral switch. For patients with critical illness the intravenous benzylpenicillin administration doses will be adjusted.
  Interventions: Drug: Penicillin
- No adjunctive treatment in combination with MRSA or MSSA or PSSA backbone therapy arm (No Intervention): No adjunctive therapy + backbone therapy arm for MRSA or MSSA or PSSA
  Participants with either MRSA or MSSA or PSSA will have no adjunctive therapy in combination with their backbone therapy arm.
- Adjunctive treatment in combination with MRSA or MSSA or PSSA backbone therapy arm (Experimental): Adjunctive therapy + backbone therapy arm for MRSA or MSSA or PSSA Intravenous clindamycin (or lincomycin) 600mg every 8 hours from platform day 1 to day 5. No dosage adjustment is needed to renal impairment.
  Interventions: Drug: Clindamycin
- Continue intravenous antibiotic therapies (backbone +/- adjunctive therapy) - standard of care arm (No Intervention): Backbone therapy arm for MRSA or MSSA or PSSA +/- adjunctive therapy will continue on intravenous antibiotic treatment for the length of time as per usual standard of care.
  Participants eligibility is assessed at Day 7 (+/- 2 days) if eligible will be randomised if not eligible then eligibility will be assess again at Day 14(+/- 2 days). If eligibility is not met at day 14 then participant is excluded from this domain.
- Switch to oral antibiotics at trial day 7 (+/- 2 days) or Day 14 (+/- 2 days) if eligible. (Experimental): Switch from intravenous backbone antibiotic for MRSA or MSSA or PSSA to oral antibiotics at the treating clinicians discretion on trial Day 7 (+/- 2 days) or trial Day 14 (+/- 2 days).
  Participants eligibility is assessed at Day 7 (+/- 2 days). If eligible will be randomised, if not eligible then eligibility will be assessed again at Day 14 (+/- 2 days). If eligibility is not met at day 14 then participant is excluded from this domain.
  Interventions: Other: Effectiveness of early switch to oral antibiotics
- No PET/CT scan - standard of care arm (No Intervention): Participants will not receive a PET/CT scan, in addition to their allocated treatment interventions.
  Participants eligibility is assessed at Day 7 (+/- 2 days) if eligible will be randomised. If eligibility is not met then participant is excluded from this domain.
- PET/CT scan at trial day 7 (+/- 2 days) if eligible (Experimental): Participant will receive a PET/CT scan at Day 5-12, in addition to their allocated treatment interventions.
  Participants eligibility is assessed at Day 7 (+/- 2 days) if eligible will be randomised. If eligibility is not met then participant is excluded from this domain.
  Interventions: Radiation: Whole body FDG PET/CT Imaging

INTERVENTIONS:
Drug: Cefazolin — Cefazolin
  Arms: Methicillin-resistant staphylococcus aureus (MRSA) - Standard + B-Lactam Arm (backbone therapy); Methicillin-susceptible staphylococcus aureus (MSSA) - Interventional Arm (backbone therapy)
Drug: Penicillin — benzylpenicillin
  Other Names: Benzylpenicillin; Penicillin G
  Arms: Penicillin-susceptible staphylococcus aureus (PSSA) - Interventional Arm (backbone therapy)
Drug: Clindamycin — Clindamycin
  Other Names: Lincomycin
  Arms: Adjunctive treatment in combination with MRSA or MSSA or PSSA backbone therapy arm
Drug: Vancomycin — Vancomycin or Daptomycin
  Other Names: Daptomycin
  Arms: Methicillin-resistant staphylococcus aureus (MRSA) - Standard + B-Lactam Arm (backbone therapy)
Other: Effectiveness of early switch to oral antibiotics — This involves testing a strategy rather than individual antibiotic agents
  Arms: Switch to oral antibiotics at trial day 7 (+/- 2 days) or Day 14 (+/- 2 days) if eligible.
Radiation: Whole body FDG PET/CT Imaging — Whole body FDG PET/CT imaging will be performed using a standardised protocol describing patient preparation and minimum specifications for radiopharmaceutical production, quality control, and PET/CT acquisition.
  Arms: PET/CT scan at trial day 7 (+/- 2 days) if eligible

SUMMARY:
The Staphylococcus aureus Network Adaptive Platform (SNAP) trial is an International Multi-Centered Randomised Adaptive Platform Clinical Trial to evaluate a range of interventions to reduce mortality for patients with Staphylococcus Aureus bacteraemia (SAB).

DETAILED DESCRIPTION:
Infection of the bloodstream with the bacterium Staphylococcus aureus (Staphylococcus aureus bacteraemia, SAB) is a serious infection that results in 15-30% of affected patients dying within three months of acquiring the infection. Treatment of this infection requires patients to be hospitalised, treated with prolonged antibiotics through an intravenous line, and carefully examined for the occurrence of complications associated with this condition. At present, there are many treatment options in current use, with no clear agreement as to which of these is best. The SNAP trial aims to identify which treatment options for SAB results in the fewest patients dying within the first 90 days after an infection.

In contrast to a conventional clinical trial, the SNAP trial will examine multiple different treatment options at once. Patients will be randomly assigned to different concurrent treatment options currently considered acceptable in routine medical care, but as the trial progresses, more patients will be assigned to treatments that appear to have better outcomes than those with worse outcomes. The trial will adapt to accumulating trial evidence, on a regular basis, by removing treatment options found to be inferior, incorporating new treatment options, and ensuring that all patients in the trial receive the best treatments once they have been identified. Over time, we hope to determine the best combination of treatment options for patients with SAB.

The SNAP Trial infrastructure will also support a number of sub-studies. A list of all active sub-studies can be found on the SNAP website: https://www.snaptrial.com.au/substudies.

ELIGIBILITY:
PLATFORM Inclusion Criteria:

Patients must fulfil all of the following criteria to be eligible to enter the SNAP trial:

1. Staphylococcus aureus complex grown from ≥1 blood culture
2. Admitted to a participating hospital at the time of eligibility assessment (OR if patient has died, they were admitted to this site anytime from the time of blood culture collection until the time of eligibility assessment)

PLATFORM Exclusion Criteria:

Potentially eligible participants meeting any of the following criteria at the time of eligibility assessment for platform entry will be excluded from the randomised platform (but may still participate in the registry):

1. Time of anticipated platform entry is greater than 72 hours post collection of the index blood culture (Where the time of culture collection is not recorded, the time of laboratory registration of the sample will be used as an alternative)
2. Polymicrobial bacteraemia, defined as more than one organism (at species level) in the index blood cultures OR in any subsequent blood culture reported between the collection of the index blood culture and platform eligibility assessment, excluding those organisms judged to be contaminants by either the microbiology laboratory or treating clinician.
3. Known previous participation in the randomised SNAP platform
4. Known positive blood culture for S. aureus (of the same silo: PSSA, MSSA or MRSA) between 72 hours and 180 days prior to the time of eligibility assessment
5. Treating team deems enrolment in the study is not in the best interest of the patient
6. Treating team believes that death is imminent and inevitable
7. Patient is for end-of-life care and antibiotic treatment is considered not appropriate
8. Patient <18 years of age and paediatric recruitment not approved at recruiting site
9. Patient has died since the collection of the index blood culture

To be included in any of the following DOMAINS the participant must met eligible for the PLATFORM (as listed above)

ADJUNCTIVE TREATMENT DOMAIN

Inclusion Criteria:

1. All participants that met the PLATFORM eligible are eligible to be included in this domain unless they meet any of the following exclusions listed.
2. Patients are eligible for this domain regardless of S. aureus susceptibility testing results to clindamycin.

Exclusion criteria:

1. Previous type 1 hypersensitivity reaction to lincosamides 2. Currently receiving clindamycin (lincomycin) or linezolid which cannot be ceased or substituted 3. Necrotising fasciitis 4. Current C. difficile associated diarrhoea (any severity) 5. Current severe diarrhoea from any cause (defined as Grade 3 or higher) 5. Known CDAD (C.Difficile Associated Diarrhoea) in the past 3 months, or CDAD relapse in the past 12 months 6. At the time of domain eligibility assessment, more than 4 hours has elapsed since platform entry 7. Treating clinician deems enrolment in this domain is not in the best interest of the patient

PSSA, MSSA TREATMENT DOMAIN (backbone)

Inclusion Criteria:

1. For PSSA silo: Index blood culture isolate is penicillin-susceptible as per the Microbiology Appendix. In short, this will require phenotypic disc testing with EUCAST (a P1 disc diffusion with zone >=26mm OR a P1 disc diffusion with zone >=26mm and the zone edge is NOT sharp) OR CLSI (a P10 disc diffusion) defined criteria.
2. For MSSA silo: Index blood culture isolate is methicillin-susceptible as per the Microbiology Appendix.

Note that where trial sites are not testing for penicillin-susceptibility, patients with MSSA/PRSA can be included in the MSSA silo, but those with MSSA/PSSA (but not confirmed with a P-disc) will be excluded from the backbone domain. The rationale for this is that patients with MSSA but not tested with a P-disc may be truly PSSA (with no blaZ). If the cefazolin inoculum effect (CIE) is a clinically relevant entity, then including patients with an organism without blaZ (and hence cannot have a CIE phenotype), will bias towards non-inferiority of cefazolin compared to (flu)cloxacillin.

For PSSA, the requirement for laboratories to use an accredited phenotypic test for a penicillin-susceptible phenotype, is to ensure clinical safety according to internationally accepted guidelines. The automated antimicrobial susceptibility testing, and other phenotypic tests, have poor sensitivity for detection of blaZ compared to a gold standard of blaZ PCR. Therefore, patients could be placed at risk of treatment with benzylpenicillin when the infecting isolate is actually blaZ positive, unless these guidelines are followed.

Exclusion Criteria (PSSA & MSSA):

1. >72 hours have elapsed since the collection of the index blood culture (i.e. the time of collection of the first positive blood culture from the patient during this episode)
2. History of type I hypersensitivity reaction (i.e. anaphylaxis or angioedema) to any penicillin or cephalosporin
3. History of severe delayed reaction (e.g. allergic interstitial nephritis, cutaneous vasculitis, Stevens-Johnson, DRESS, etc.) to any penicillin or cephalosporin
4. PSSA silo: Non-severe rash to any penicillin (unless patient has been subsequently de-labelled; this criteria does not include criteria 2 and 3 above), or MSSA silo: Non-severe rash to cefazolin or any penicillin (unless patient has been subsequently de-labelled); (Nausea, diarrhoea, headache, and other non-specific symptoms are NOT allergies, they are drug intolerance, and they are not exclusion criteria. Similarly, a vague history of an allergy of unclear nature, or a family history of allergy are not exclusions.)
5. Treating team deems enrolment in this domain is not in the best interest of the patient
6. Currently receiving maintenance dialysis (haemodialysis or peritoneal dialysis); (Acute renal replacement therapy (including CRRT, haemodialysis or peritoneal dialysis) are not exclusions. Such patients are eligible as long as appropriate vascular access is available or can be arranged.)
7. Polymicrobial bacteraemia (defined as more than one organism [at species level] in blood cultures, excluding those organisms judged to be contaminants by either the microbiology laboratory or treating clinician) reported between collection of the index blood culture and backbone domain eligibility assessment
8. Patient currently being treated with a systemic antibacterial agent that cannot be ceased or substituted for interventions allocated within the platform (unless antibiotic is listed in Table 1 of the DSA, which specifies allowed antibiotics with limited absorption from the gastrointestinal tract or negligible antimicrobial activity against S. aureus)

MRSA TREATMENT DOMAIN (backbone)

Inclusion Criteria:

1. MRSA confirmed microbiologically

Exclusion Criteria:

1. Time to allocation reveal is >72 hours from time of index blood culture collection
2. Severe allergy to any beta-lactam (including cefazolin) Immediate severe allergy: Anaphylaxis/angioedema Severe delayed allergy: Severe cutaneous adverse reaction (SCAR; including Steven Johnson Syndrome, Toxic Epidermal Necrolysis, Drug Rash with Eosinophilia and Systemic Symptoms (DRESS) and acute generalised exanthematous pustulosis (AGEP)), severe drug induced liver injury, proven allergic interstitial nephritis, immune-mediated haemolytic anaemia and other severe cytopenia.
3. Non-severe rash to cefazolin Nausea, diarrhoea, headache and other non-specific symptoms are NOT allergies, they are drug intolerance, and they are not exclusion criteria. Similarly, a vague history of an allergy of unclear nature, or a family history of allergy are not exclusions.)

3. Severe allergy or non-severe rash to both vancomycin AND daptomycin Vancomycin infusion reaction (formerly known as "red man syndrome") is due to direct histamine release and is not generally an allergy, and therefore is not considered an exclusion.

5. Treating team deems enrolment in the domain is not in the best interest of the patient 6. Polymicrobial bacteraemia (defined as more than one organism [at species level] in blood cultures, excluding those organisms judged to be contaminants by either the microbiology laboratory or treating clinician) reported between collection of the index blood culture and backbone domain eligibility assessment.

7. Patient currently being treated with a systemic antibacterial agent that cannot be ceased or substituted for interventions allocated within the platform (unless antibiotic is listed in Table 1 of the DSA, which specifies allowed antibiotics with limited absorption from the gastrointestinal tract or negligible antimicrobial activity against S. aureus)

EARLY ORAL SWITCH DOMAIN

Inclusion Criteria:

Day 7 (+/- 2 days):

1. Clearance of SAB by platform Day 2: blood cultures negative for S. aureus from platform Day 2 onwards AND no known subsequent positive blood cultures
2. Afebrile (<37.8°C) for the past 72 hours (at time of judging eligibility)
3. Primary focus is either line related (either central or peripheral IV cannula) or skin and soft tissue, AND source control achieved (for 'line-related' this means line removed; for 'skin and soft tissue' means site PI considers source control to have been achieved and any abscess more than 2cm diameter has been drained)
4. No evidence of metastatic foci (on clinical or radiological examination, but radiological imaging is not required to exclude metastatic foci if not clinically indicated)

Day 14 (+/- 2 days):

1. Clearance of SAB by platform Day 5: blood cultures negative for S. aureus from platform Day 5 (+/-1 day) AND no known subsequent positive blood cultures. If the most recent blood culture from Day 2-4 is negative for S. aureus, blood cultures do not need to be repeated on Day 5 to fulfil eligibility criteria (Day 5 blood cultures will be assumed to be negative in this situation)
2. Afebrile (<37.8°C) for the past 72 hours (at time of judging eligibility)
3. Site Principal Investigator has determined that source control is adequate

Exclusion Criteria:

When judging eligibility at platform Day 7 (+/- 2 days) and at Day 14 (+/- 2 days), exclusion criteria are:

1. Adherence to oral agents unlikely (as judged by site PI in consultation with the treating team)
2. Unreliable gastrointestinal absorption (e.g. vomiting, diarrhoea, nil by mouth, anatomical reasons)
3. There are no appropriate oral antibiotics due to contraindications, drug availability, or antibiotic resistance
4. Ongoing IV therapy unsuitable e.g. no IV access
5. Clinician deems not appropriate for early oral switch
6. Patient no longer willing to participate in domain In the lead-up to judging eligibility, it may be helpful to discuss with the patient the potential for continued IV treatment versus oral switch, to allow hospital discharge planning
7. Clinical team deems that sufficient duration of antibiotic therapy has already been provided

Exclusions when judging eligibility for early oral switch at trial Day 7 (+/- 2 days):

1. Presence of prosthetic cardiac valve, pacemaker or other intracardiac implant
2. Presence of intravascular clot, graft, or other intravascular prosthetic material Intravascular clot excludes superficial peripheral IV line-related thrombophlebitis. Intravascular prosthetic material excludes coronary artery stents)
3. Intravascular/intracardiac infections (e.g. endocarditis, mycotic aneurysm)
4. Presence of other intracardiac abnormalities felt to put patient at increased risk of endocarditis (e.g., bicuspid aortic valve)

PET/CT DOMAIN

Inclusion Criteria:

1. PET/CT participating site
2. Patient is accessible for PET/CT - a patient is considered accessible if the site team are able to access the participant medical records, arrange for a PET/CT scan for the patient, and discuss this domain with the patient and their treating healthcare providers.

Exclusion Criteria:

1. Pregnant - patients of childbearing potential should be assessed for pregnancy status and a pregnancy test performed (if not performed within the past 10 days)
2. Currently breastfeeding
3. < 18 years of age
4. Patient has had PET/CT in the past 7 days
5. Patient needs PET/CT in the next 7 days (in the opinion of the clinical team, at the time of eligibility assessment)
6. Clinically unstable for PET/CT (as judged by the treating clinical team, taking into account need for organ support (including inotropes) and capacity to lie flat for the PET/CT)
7. Contraindication to PET/CT (e.g., claustrophobia, persistently elevated blood sugar levels [>12.5mmol/L] that cannot be corrected).
8. Patient no longer willing to participate in the domain - in the days leading up to judging eligibility, it may be helpful to discuss with the patient the potential for PET/CT vs no PET/CT to allow imaging planning
9. Clinician deems participation in this domain is not in the patient's best interests

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 90 days after platform entry | From randomisation (day 1) until day 90
  The primary endpoint for all cells and domains will be all-cause mortality at 90 days after platform entry.
  The primary endpoint will be determined through a search of hospital databases for a record of a participant's death, or follow-up contact with the participant's community healthcare provider, or follow-up contact with the patient or their nominated carer, or linkage with death registries.

SECONDARY OUTCOMES:
Core1: All-cause mortality at 14, 28 and 42 days after platform entry | From randomisation (day 1) until day 14, 28, and 42
  Determined through a search of hospital databases for a record of a participant's death, or follow-up contact with the participant's community healthcare provider, or follow-up contact with the patient or their nominated carer, or linkage with death registries.
Core2: Duration of survival censored at 90 days after platform entry | From randomisation (day 1) until day 90
  Determined through a search of hospital databases for a record of a participant's death, or follow-up contact with the participant's community healthcare provider, or follow-up contact with the patient or their nominated carer, or linkage with death registries.
Core3: Length of stay of acute index inpatient hospitalisation for those surviving until discharge from acute inpatient facilities (excluding HITH/COPAT/OPAT/rehab). | From randomisation (day 1) until discharge from acute inpatient facilities, truncated at 90 days.
  Acute index hospitalisation is defined as continuous hospital admission to one or more acute inpatient facilities for the index episode. This does not include HITH/OPAT/COPAT and stepdown inpatient rehabilitation/post-acute care. It does include admission to acute care hospitals immediately preceding and following those at the enrolling site.
Core4: Length of stay of total index hospitalisation for those surviving until hospital discharge (including HITH/COPAT/OPAT/rehab) | From randomisation (day 1) to discharge from total index hospitalisation, truncated at 90 days
  Total index hospitalisation is defined as continuous hospital admission to one or more inpatient facilities for the index episode, including HITH/OPAT/COPAT and stepdown inpatient rehabilitation/post-acute care (if continuous with the initial inpatient admission).
  It includes admission to acute care hospitals immediately preceding and following those at the enrolling site.
Core5: Time to being discharged alive from the total index hospitalisation (including HITH/COPAT/OPAT/rehab) truncated at 90 days after platform entry | From randomisation (day 1) to discharge from total index hospitalisation, truncated at 90 days
  and all deaths within 90 days will be considered '90 days'
Core6: Microbiological treatment failure defined as positive sterile site culture for S. aureus [of the same silo as the index isolate between 14 and 90 days after platform entry). | From day 14 until day 90
  A sterile site means any sites deep to the skin and skin structures, including deep visceral and musculoskeletal abscesses that have been obtained in a sterile manner.
Core7: Diagnosis of new foci between 14 and 90 days after platform entry. | From day 14 until day 90
  The presence of new foci will be determined by the site investigator and can incorporate clinical, radiological, microbiological and pathological findings.
Core8: C. difficile diarrhoea as determined by a clinical laboratory in the 90 days following platform entry for participants ≥2 years of age. | From randomisation (day 1) until day 90
  This means a stool submitted to a clinical laboratory has tested positive for C. difficile toxin or toxin gene.
Core9: Serious adverse reactions (SARs) in the 90 days following platform entry | From randomisation (day 1) until day 90
  SARs defined only as serious events that are attributable to one or more randomised study interventions
Core10: Health economic costs as detailed in the health ecnomics appendix. | From randomisation (day 1) until day 90
  Including hospital length of stay, readmissions, and patient employment status.
Core11: Proportion of participants who have returned to their usual level of function at day 90. | From randomisation (day 1) until day 90
  Determined by whether the modified functional bloodstream infection score (FBIS) remained the same or improved between baseline and 90 days after platform entry where baseline=best score within the 4 weeks prior to platform entry.
Core12: Desirability of outcome ranking 1 (DOOR1; modified Antibiotic Resistance Leadership Group version) | From randomisation (day 1) until day 90
  See Core Protocol; unable to insert DOOR1 table
Core13: Desirability of outcome ranking 2 (DOOR2; SNAP version) | From randomisation (day 1) until day 90
  See Core Protocol; unable to insert DOOR2 table
Core14: Total number of antibiotic days (IV and/or oral/enteral) in the 90 days following platform entry. | From randomisation (day 1) until day 90
  All antibiotics should be included, not only those intended for treatment of S. aureus bacteraemia. It also includes prophylactic dose antibiotics (e.g., prophylactic dose trimethoprim-sulfamethoxazole).
  All days on which any antibiotic dose is received should be counted - i.e. we are counting the number of whole or part days on which any antibiotics are received (not the number of defined daily doses of antibiotics).
  Topical, inhaled or other routes of administration besides IV or oral/enteral should not be counted.
Core15: Days alive and free of antibiotics in the 90 days following platform entry. | From randomisation (day 1) until day 90
  All antibiotics should be included, not only those intended for treatment of S. aureus bacteraemia. It also includes prophylactic dose antibiotics (e.g., prophylactic dose trimethoprim-sulfamethoxazole).
  All days on which any antibiotic dose is received should be counted - i.e. we are counting the number of whole or part days on which any antibiotics are received (not the number of defined daily doses of antibiotics).
  Topical, inhaled or other routes of administration besides IV or oral/enteral should not be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Steven Tong, Study Chair — University of Melbourne / Melbourne Health; Prof Joshua Davies, Study Chair — Menzies School of Research / Hunter New England Medical Centre
Locations (151):
- Houston Methodist Research Institute, Houston, Texas, United States
- Australia (51):
  - Canberra Hospital, Garran, Australia Capital Territory
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation and General Hospital, Concord, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - John Hunter Children's Hospital, Newcastle, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Ipswich Hospital, Ipswich, Queensland
  - Logan Hospital, Meadowbrook, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Robina Hospital, Robina, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Lyell McEwin Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Women and Children's Hospital, North Adelaide, South Australia
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston Hospital, Launceston, Tasmania
  - Grampians Health, Ballarat, Victoria
  - Bendigo Health, Bendigo, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Children's Hospital, Clayton, Victoria
  - Monash Health - Monash Medical Centre & Jesse McPherson Private Hospital, Clayton, Victoria
  - Western Health - Footscray, Joan Kirner & Sunshine Hospitals, Footscray, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Barwon Health - University Hospital Geelong, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Children's Hospital Melbourne, Parkville, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - La Trobe Regional Hospital, Traralgon, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Perth Children's Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Armadale Hospital, Perth, Western Australia
- Canada (37):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Center, Calgary, Alberta
  - Rockyview Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Richmond Hospital, Richmond, British Columbia
  - Fraser Health Authority - Surrey Memorial Hospital, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Grace Hospital, Winnipeg, Manitoba
  - Eastern Health - Health Sciences Centre (Memorial University), St. John's, Newfoundland and Labrador
  - Eastern Regional Health Authority - St. Clare's Mercy Hospital, St. John's, Newfoundland and Labrador
  - Toronto East Health Network - Michael Garron Hospital, East York, Ontario
  - University Health Network - Toronto General Hospital, East York, Ontario
  - Hamilton Health Sciences - Hamilton General Hospital, Hamilton, Ontario
  - Hamilton Health Sciences - Juravinski Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre - University Hospital, LHSC, London, Ontario
  - Niagara Health - Niagara Falls Site, Niagara Falls, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Niagara Health - St. Catharines Site, St. Catharines, Ontario
  - Unity Health - St Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Sinai Heath System - Mount Sinai Hospital, Toronto, Ontario
  - Unity Health Toronto - St Joseph's Health Centre, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
  - CISSS - Hôpital Cité-de-la-Santé Hospital, Laval, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre - Montral General Hospital, Montreal, Quebec
  - McGill University Health Centre - Montreal Children's Hospital, Montreal, Quebec
  - McGill University Health Centre - Royal Victoria Hospital, Montreal, Quebec
  - Hôpital Régional de Saint Jérôme, Saint-Jérôme, Quebec
  - University of Sherbrooke Health Centre - Hospital Fleurimont, Sherbrooke, Quebec
  - University of Sherbrooke Health Centre - Hotel Dieu, Sherbrooke, Quebec
- Israel (4):
  - Rambam Health Care Campus, Haifa, Haifa District
  - Beilinson Hospital, Petah Tikva, Petah Tikva
  - Schneider Hospital, Petah Tikva
  - Sheba Medical Centre, Ramat Gan
- Science Tokyo University Hospital, Ichikawa, Chiba, Japan
- Netherlands (6):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - UMC Groningen, Groningen
  - Antonius Ziekenhuis, Nieuwegein
  - Radboud University Medical Center, Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
  - University Medical Center Utrecht, Utrecht
- New Zealand (11):
  - Auckland City Hospital, Grafton, Auckland
  - Middlemore Hospital, Otahuhu, Auckland
  - North Shore Hospital, Takapuna, Auckland
  - Christchurch Hospital, Christchurch, Canterbury
  - Waikato Hospital, Hamilton, Hamilton
  - Hutt Valley Hospital, Boulcott, Lower Hutt
  - Tauranga Hospital, Tauranga, Tauranga
  - Wellington Hospital, Newtown, Wellington Region
  - Whangarei Hospital, Whangarei, Whangarei
  - Starship Hospital, Auckland
  - KidzFirst, Auckland
- Singapore (3):
  - National University Hospital, Singapore, Singapore
  - Singapore General Hospital, Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore, Singapore
- South Africa (3):
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg
  - Helen Joseph Hospital, Johannesburg
  - Rahima Moosa Mother and Child Hospital, Johannesburg
- United Kingdom (34):
  - NHS Grampian, Aberdeen
  - University Hospitals Birmingham, Birmingham
  - Brighton and Sussex University Hospitals, Brighton
  - North Bristol, Bristol
  - University Hospitals Bristol and Weston, Bristol
  - Cambridge University Hospitals, Cambridge
  - Cardiff and Vale University, Cardiff
  - Royal Cornwall Hospitals, Cornwall
  - Royal Devon University Healthcare, Devon
  - NHS Tayside, Dundee
  - Lothian Western General, Edinburgh
  - Greater Glasgow and Clyde, Glasgow
  - NHS Golden Jubilee, Glasgow
  - Hull University Teaching Hospitals, Hull
  - Leeds Teaching Hospitals, Leeds
  - Liverpool University Hospital, Liverpool
  - Barts Health, London
  - Great Ormond Street, London
  - Guys and St Thomas', London
  - Imperial College Healthcare, London
  - Kings College Hospital, London
  - Royal Free London, London
  - University College London Hospitals, London
  - Whittington Health, London
  - Manchester University Hospitals, Manchester
  - Newcastle Upon Tyne Hospitals, Newcastle upon Tyne
  - Nottingham University Hospitals, Nottingham
  - Oxford University Hospitals, Oxford
  - Sheffield Teaching Hospitals, Sheffield
  - South Tees Hospitals, South Tees
  - University Hospital Southampton, Southampton
  - NHS Forth Valley, Stirling
  - University Hospitals of North Midlands, Stoke
  - Swansea Bay University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting information will be available 12 months after the publication of the primary results manuscript and will be available for a 10 year period.
Access Criteria: • All requests for data sharing must be accompanied by a SNAP data access request from, a study proposal with clear statement of aims and hypotheses, and a statistical analysis plan. All applications will be assessed by the SNAP Trial Steering Committee. Applications from investigators with suitable academic capability to conduct the proposed work will be given consideration. If a proposal is approved, a signed data transfer agreement will be required before data sharing.
URL: https://www.snaptrial.com.au/for-investigators#integrity

REFERENCES:
- [Background] Tong SYC, Mora J, Bowen AC, Cheng MP, Daneman N, Goodman AL, Heriot GS, Lee TC, Lewis RJ, Lye DC, Mahar RK, Marsh J, McGlothlin A, McQuilten Z, Morpeth SC, Paterson DL, Price DJ, Roberts JA, Robinson JO, van Hal SJ, Walls G, Webb SA, Whiteway L, Yahav D, Davis JS; Staphylococcus aureus Network Adaptive Platform (SNAP) Study Group. The Staphylococcus aureus Network Adaptive Platform Trial Protocol: New Tools for an Old Foe. Clin Infect Dis. 2022 Nov 30;75(11):2027-2034. doi: 10.1093/cid/ciac476. PMID 35717634
- [Background] Sakai K, Homma H, Lee JA, Fukushima T, Santa T, Tashiro K, Iwatsubo T, Imai K. Emergence of D-aspartic acid in the differentiating neurons of the rat central nervous system. Brain Res. 1998 Oct 12;808(1):65-71. doi: 10.1016/s0006-8993(98)00599-x. PMID 9795139
- [Background] Mayer EA. Clinical implications of visceral hyperalgesia. Contemp Intern Med. 1994 Jul;6(7):42-54. PMID 10150304
- [Background] Pryce W. Have skills, will travel. Nurs Times. 1999 Mar 24-30;95(12):26. No abstract available. PMID 10232234
- [Background] de Kretser D, Mora J, Bloomfield M, Campbell A, Cheng MP, Guy S, Hensgens M, Kalimuddin S, Lee TC, Legg A, Mahar RK, Marks M, Marsh J, McGlothin A, Morpeth SC, Sud A, Ten Oever J, Yahav D, Bonten M, Bowen AC, Daneman N, van Hal SJ, Heriot GS, Lewis RJ, Lye DC, McQuilten Z, Paterson DL, Owen Robinson J, Roberts JA, Scarborough M, Webb SA, Whiteway L, Tong SYC, Davis JS, Walls G, Goodman AL; SNAP Early Oral Switch Domain-Specific Working Group and SNAP Global Trial Steering Committee; SNAP Trial Group. Early Oral Antibiotic Switch in Staphylococcus aureus Bacteraemia: The Staphylococcus aureus Network Adaptive Platform (SNAP) Trial Early Oral Switch Protocol. Clin Infect Dis. 2024 Oct 15;79(4):871-887. doi: 10.1093/cid/ciad666. PMID 37921609
- [Background] Yamanaka T, Him A, Cameron SA, Dutia MB. Rapid compensatory changes in GABA receptor efficacy in rat vestibular neurones after unilateral labyrinthectomy. J Physiol. 2000 Mar 1;523 Pt 2(Pt 2):413-24. doi: 10.1111/j.1469-7793.2000.t01-1-00413.x. PMID 10699085
- [Derived] Mahar RK, McGlothlin A, Dymock M, Barina L, Bonten M, Bowen A, Cheng MP, Daneman N, Goodman AL, Lee TC, Lewis RJ, Lumley T, McLean ARD, McQuilten Z, Mora J, Paterson DL, Price DJ, Roberts J, Snelling T, Tverring J, Webb SA, Yahav D, Davis JS, Tong SYC, Marsh JA; SNAP Global Trial Steering Committee. Statistical documentation for multi-disease, multi-domain platform trials: our experience with the Staphylococcus aureus Network Adaptive Platform trial. Trials. 2025 Feb 11;26(1):49. doi: 10.1186/s13063-024-08684-8. PMID 39934879
- [Derived] Mahar RK, McGlothlin A, Dymock M, Lee TC, Lewis RJ, Lumley T, Mora J, Price DJ, Saville BR, Snelling T, Turner R, Webb SA, Davis JS, Tong SYC, Marsh JA; SNAP Global Trial Steering Committee. A blueprint for a multi-disease, multi-domain Bayesian adaptive platform trial incorporating adult and paediatric subgroups: the Staphylococcus aureus Network Adaptive Platform trial. Trials. 2023 Dec 6;24(1):795. doi: 10.1186/s13063-023-07718-x. PMID 38057927
- See also: SNAP Trial Website — http://www.snaptrial.com.au/